CLINICAL TRIAL: NCT06975085
Title: Understanding and Addressing Rejection of Personalized Breast Cancer Risk Information in Women
Brief Title: Understanding and Addressing Rejection of Personalized Breast Cancer Risk Information: Administrative Supplement Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0345; R01CA279953 (NIH)
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Female
Keywords: breast cancer risk; risk perceptions; screening intentions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer risk presentation (Other): All participants are presented with their personal breast cancer risk, estimated using the Gail Model
  Interventions: Behavioral: Presentation of a personal breast cancer risk estimate

INTERVENTIONS:
Behavioral: Presentation of a personal breast cancer risk estimate — Participants answer questions that are used to calculate their personal breast cancer risk using the Gail Model. This risk estimate is presented to participants using written text and an icon array.

SUMMARY:
The Understanding and Addressing Rejection of Personalized Cancer Risk Information study is a longitudinal study conducted to understand the nature of phenomenon of personalized cancer risk rejection in the context of mammography screening.

DETAILED DESCRIPTION:
The Understanding and Addressing Rejection of Personalized Cancer Risk Information study seeks to understand the nature of the phenomenon of personalized cancer risk rejection in the context of mammography screening by testing hypotheses about why women reject their risk estimate and the influence of rejection on screening intentions.

The Breast Cancer Risk Assessment Tool (BCRAT) will be used to asses participant's breast cancer risk. This model is designed to estimate breast cancer risk in women 35-84, and uses the following predictors: 1) age, 2) age at first menstrual period, 3) age at first live birth, 4) first-degree relatives with breast cancer, 5) previous breast biopsy with atypical hyperplasia, and 6) race/ethnicity. Participants will be required to complete a survey in which they receive their BCRAT model risk estimate and respond to that risk estimate.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Age 39-74 (i.e., people who are eligible for routine breast cancer screening and for whom guidelines recommend an informed, risk-based decision)
3. English literacy
4. Black or African American race

Exclusion Criteria:

1. Prior diagnosis of

1. breast cancer
2. Ductal carcinoma in situ (DCIS)
3. Lobular carcinoma in situ (LCIS)
4. Known BRCA1/2 gene mutation
5. Cowan syndrome
6. Li-Fraumeni syndrome
7. Having received previous chest radiation for treatment of Hodgkin's lymphoma.

Ages: 39 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Risk rejection as measured by a numeric estimate | at baseline survey
  Participants are asked whether they agree or disagree with their Gail Model risk estimate. An open text box allows them to write the risk number that they believe is accurate for them.
Risk-concordant information seeking | at baseline survey
  Participants will be given the opportunity to get more information about breast cancer screening, and will be given response options to receive information for women at lower than average risk, higher than average risk, or women with risk that is "about the same as a typical woman". Concordance is measured by agreement between the participants' actual risk estimate and the option that they choose.
Screening intentions | at baseline survey
  Participants are asked: In the next 12 months, do you plan to get a mammogram? The question is answered on a 5-point will-will not Likert scale. 1=definitely will not, 2=probably will not, 3=maybe, 4=probably will, 5=definitely will

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Scherer, PhD, Principal Investigator — University of Colorado, Denver; Erika Waters, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the protocol, code books, and data set associated with this study on the Open Science Framework after ensuring that it is completely anonymized.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting information will be made available when we submit the first manuscript to a journal for review.
Access Criteria: Anyone will be able to access the IPD and supporting information by downloading it from OSF.
URL: https://osf.io